CLINICAL TRIAL: NCT00169533
Title: An Open Label, Phase 1b Rollover Study to Assess the Long-Term Safety Profile of Lapatinib (GW572016) in Cancer Patients.
Brief Title: Rollover Study Of Lapatinib In Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EGF19060
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Neoplasms, Breast
Keywords: safety; tolerating lapatinib; Lapatinib
MeSH Terms: conditions — Breast Neoplasms | interventions — Lapatinib

ARMS (1):
- Arm 1 (Experimental): Lapatinib either 750, 1000, 1250 or 1500 mgs
  Interventions: Drug: GW572016 oral tablets

INTERVENTIONS:
Drug: GW572016 oral tablets — Lapatinib either at 750, 1000, 1250 or 1500 mgs

SUMMARY:
The EGF19060 study is a rollover study to evaluate the long term safety of lapatinib and to provide lapatinib to patients who had a positive response in previous lapatinib studies until lapatinib is available pending FDA approval.

ELIGIBILITY:
Inclusion Criteria:

* Currently receiving clinical benefit as defined by CR, PR or SD from treatment with lapatinib through participation in a Phase I study of lapatinib either as monotherapy or as part of a combination regimen.
* Ability to understand and provide written informed consent to participate in this trial.
* Is male or female.
* Female and male subjects agree to the protocol specific birth control measures

Exclusion Criteria:

* Permanent discontinuation of lapatinib in the previous study due to intolerance or treatment failure.
* Is a pregnant or lactating female.
* Is considered medically unfit for the study by the investigator as a result of the medical interview, physical exam, or screening investigations.
* Currently receiving treatment with any medications listed on the prohibited medication list (see Section 7.2).
* Has Class III or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system.
* Has a left ventricular ejection fraction (LVEF) < 40% based on MUGA or ECHO.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2004-08-19 (Actual); Primary Completion 2009-05-05 (Actual); Study Completion 2009-05-05 (Actual)

PRIMARY OUTCOMES:
To determine the long-term safety and tolerability of lapatinib as monotherapy or in combination regimen | Ongoing study until the new lapatinib rollover study, EGF111767, is approved at the current sites.

SECONDARY OUTCOMES:
Assess the Long-Term Safety Profile of Lapatinib (GW572016) in Cancer Patients, Overall survival | Ongoing study until the new lapatinib rollover study, EGF111767, is approved at the current sites.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (12):
- United States (10):
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Lebanon, New Hampshire
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, San Antonio, Texas
- GSK Investigational Site, Edmonton, Alberta, Canada
- GSK Investigational Site, Tel Aviv, Israel

REFERENCES:
- See also: Results for study EGF19060 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/EGF19060?search=study&search_terms=EGF19060#rs